CLINICAL TRIAL: NCT02129829
Title: Prevention of Liver Fibrosis and Cancer in Africa. Observational Study of Screening, Assessment and Treatment for Chronic Hepatitis B Virus Infection
Brief Title: PROLIFICA - West African Treatment Cohort for Hepatitis B
Acronym: WATCH
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Department of State for Health and Social Welfare, The Gambia (Other Government); UFR Sante de Thies, Senegal (Unknown); Cheikh Anta Diop University, Senegal (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: WMDH-P34114
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Hepatitis B, Chronic; Hepatocellular Carcinoma
Keywords: Cirrhosis; HBV; HIV; HCV
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular; Fibrosis | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, urine and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observational Group: Patients whose viral load, ALT value and fibrosis status does not meet EASL criteria for treatment and are observed 6 monthly
- Treatment Group (Tenofovir disoproxil): Patients who meet EASL treatment criteria who receive Tenofovir disoproxil
  Interventions: Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Tenofovir disoproxil — Tenofovir disoproxil 245 mg once daily
  Other Names: Viread
  Groups: Treatment Group (Tenofovir disoproxil)

SUMMARY:
The West African Treatment Cohort for Hepatitis B (WATCH) study is a component of the European Commission Funded FP7 project PROLIFICA. It aims to evaluate a number of steps required to successfully treat patients with chronic hepatitis B virus infection to prevent cirrhosis and liver cancer. The first step is to determine whether screening for hepatitis B using a point of care test is feasible and effective. The second is to monitor linkage from screening into care. The third is to evaluate cheap non-invasive assessments to determine the need for treatment. The fourth is to determine what proportion of patients meet treatment eligibility criteria. The fifth step is to establish a treatment cohort which can be used to measure adherence to therapy and avoidance of HBV related complications. A parallel untreated cohort will be established to determine whether treatment criteria are relevant in this West African setting by monitoring for complications of HBV infection.

DETAILED DESCRIPTION:
Objectives Primary:

To determine whether suppression of HBV with a nucleotide analogue reduces the risk of liver cancer in West African populations.

Secondary:

To demonstrate that HBV replication can be effectively suppressed with a nucleotide analogue in West African populations To evaluate whether European treatment guidelines are applicable in West Africa To establish the applicability and efficacy of population based screening, clinical assessment and treatment in West Africa To enumerate the proportion of the adult population who carry HBV To evaluate the proportion of the HBV infected population who meet European Association for Study of the Liver (EASL) criteria for treatment

Endpoints Primary:

Incidence of Hepatocellular Carcinoma over the period of study in a treated cohort of patients with chronic HBV compared to historical controls

Secondary:

Proportion of adult population in Gambia and Senegal with chronic HBV infection Proportion of patients with chronic HBV infection who meet EASL treatment criteria Proportion of patients with undetectable HBV DNA < 400 copies/ml at 1, 2, 3, 4 and 5 years of treatment.

Incidence of hepatocellular Carcinoma in patients who do not meet EASL treatment criteria.

Treatment adherence rate. Average change in Fibroscan score after 3 and 5 years of treatment Emergence of resistance to treatment

Study Phase 4

Study Design A two part study:

Part 1 - Population based screening for HBV infection using a point-of-care test.

Part 2 - Non-randomised, open label, treatment cohort with parallel observation cohort

Number of Subjects Part 1:

Approximately 13,500 adults from the general population.

Part 2:

300 subjects in the treatment group 600 subjects in the observation group

Study Population Part 1:

Males and females aged over 30 years

Part 2:

Patients with chronic hepatitis B virus infection identified through population based screening.

Treatment Cohort There will be a single treatment group of 300 patients who meet EASL treatment criteria.

Schedule of Study Visits Part 1:

A single visit to an individual at their home or workplace when screening for HBV infection will be performed using a point-of-care test..

Part 2:

One screening visit will be performed to determine viral load, liver function tests, clinical examination, ultrasound examination and liver fibrosis assessment.

A second visit, 1 - 3 months later, will be used to verify viral load and ALT values

For those on treatment cohort:

A baseline visit will take place 2 weeks after the second screening visit and study drug will be dispensed with instructions for the patient.

First follow-up will be at 1 month to check adherence Second follow-up will be at 3 months for viral load and liver functions tests Treatment subjects will be seen every 3 months to dispense study drug and check compliance Viral load, liver function, renal function, AFP and ultrasound will be performed every 6 months.

Serum/plasma and urine samples for biomarkers of cancer development will be taken at baseline and annually.

Population Screening (Part 1 only) Communities will be sensitised about the study prior to visits by fieldworkers to individual homes, places of work or recreational facilities. A point-of-care test based on the detection of hepatitis B surface antigen (HBsAg) in a finger-prick blood sample will be used for screening. Subjects with a positive test will be given a hospital appointment for full clinical assessment.

Efficacy Evaluations (Part 2 only) Detection of liver cancer - Surveillance for liver cancer will be made using ultrasound and serum AFP every 6 months on all subjects. In some centres further imaging will be available.

Liver cancer will be diagnosed according to the following criteria:

* Liver mass with typical features of hepatocellular carcinoma on two imaging modalities (ultrasound, bubble ultrasound or CT), or
* liver mass on ultrasound and AFP > 400 iu/ml or
* histological or cytological confirmation of diagnosis.

Viral Load - viral load will be measure on EDTA plasma samples using an in-house real-time PCR assay verified for accuracy against commercial assays every 6 months.

Safety Evaluations (Part 2 only) Liver function tests, serum phosphate and renal function will be tested every 6 months

Evaluation of treatment guidelines Subjects who do not meet the EASL treatment criteria at baseline will be enrolled in the observational study with surveillance for liver cancer every 6 months

Detection of viral resistance Viral load monitoring of patients in the treatment study every 6 months will be used to detect possible virological resistance. A rise in viral load from nadir values or reappearance of detectable viraemia in patients who had achieved undetectable viral load will be investigated for emergence of viral sequence variants and for adherence to therapy

ELIGIBILITY:
Inclusion Criteria:

* Adult Informed consent HBsAg positive Resident in Gambia or Senegal

Exclusion Criteria:

* HIV infection HCV infection Known liver cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults are included for community screening. Selection criteria (below) are applied for recruitment into cohorts
Sampling Method: Probability Sample
Enrollment: 1079 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of HCC or decompensated cirrhosis | 5 years
  Subjects will be reviewed 6 monthly with liver biochemistry and ultrasound to detect onset of hepatocellular carcinoma or decompensated cirrhosis

SECONDARY OUTCOMES:
Uptake of screening | 2 years
  Proportion of community subjects who accept screening tests
Prevalence of HBV infection | 2 years
  Proportion of patients who test positive for HBsAg
Rate of linkage into care | 2 years
  Proportion of patients who test positive for HBsAg who attend clinic for assessment
Treatment rate | 2 years
  Proportion of patients with HBsAg who meet EASL treatment criteria

OTHER OUTCOMES:
Reliability of PoC test | 2 years
  Sensitivity and specificity of capillary blood sample HBsAg test applied at point of care
Accuracy of non-invasive fibrosis assessment | 2 years
  Sensitivity, specificity and ROC analysis of Fibroscan, APRI and FIB4 tests compared to liver biopsy to assess liver fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thursz, MD FRCP, Principal Investigator — Imperial College London
Locations (2):
- UFR Sante Thies,, Thiès, Senegal
- MRC Laboratories Hospital, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemoine M, Shimakawa Y, Njie R, Njai HF, Nayagam S, Khalil M, Goldin R, Ingiliz P, Taal M, Nyan O, Corrah T, D'Alessandro U, Thursz M. Food intake increases liver stiffness measurements and hampers reliable values in patients with chronic hepatitis B and healthy controls: the PROLIFICA experience in The Gambia. Aliment Pharmacol Ther. 2014 Jan;39(2):188-96. doi: 10.1111/apt.12561. Epub 2013 Dec 5. PMID 24308698
- [Background] Lemoine M, Shimakawa Y, Njie R, Taal M, Ndow G, Chemin I, Ghosh S, Njai HF, Jeng A, Sow A, Toure-Kane C, Mboup S, Suso P, Tamba S, Jatta A, Sarr L, Kambi A, Stanger W, Nayagam S, Howell J, Mpabanzi L, Nyan O, Corrah T, Whittle H, Taylor-Robinson SD, D'Alessandro U, Mendy M, Thursz MR; PROLIFICA investigators. Acceptability and feasibility of a screen-and-treat programme for hepatitis B virus infection in The Gambia: the Prevention of Liver Fibrosis and Cancer in Africa (PROLIFICA) study. Lancet Glob Health. 2016 Aug;4(8):e559-67. doi: 10.1016/S2214-109X(16)30130-9. PMID 27443781
- [Background] Nayagam S, Conteh L, Sicuri E, Shimakawa Y, Suso P, Tamba S, Njie R, Njai H, Lemoine M, Hallett TB, Thursz M. Cost-effectiveness of community-based screening and treatment for chronic hepatitis B in The Gambia: an economic modelling analysis. Lancet Glob Health. 2016 Aug;4(8):e568-78. doi: 10.1016/S2214-109X(16)30101-2. PMID 27443782
- [Background] Shimakawa Y, Ndow G, Njie R, Njai HF, Takahashi K, Akbar SMF, Cohen D, Nayagam S, Jeng A, Ceesay A, Sanneh B, Baldeh I, Imaizumi M, Moriyama K, Aoyagi K, D'Alessandro U, Mishiro S, Chemin I, Mendy M, Thursz MR, Lemoine M. Hepatitis B Core-related Antigen: An Alternative to Hepatitis B Virus DNA to Assess Treatment Eligibility in Africa. Clin Infect Dis. 2020 Mar 17;70(7):1442-1452. doi: 10.1093/cid/ciz412. PMID 31102406
- [Background] Shimakawa Y, Njie R, Ndow G, Vray M, Mbaye PS, Bonnard P, Sombie R, Nana J, Leroy V, Bottero J, Ingiliz P, Post G, Sanneh B, Baldeh I, Suso P, Ceesay A, Jeng A, Njai HF, Nayagam S, D'Alessandro U, Chemin I, Mendy M, Thursz M, Lemoine M. Development of a simple score based on HBeAg and ALT for selecting patients for HBV treatment in Africa. J Hepatol. 2018 Oct;69(4):776-784. doi: 10.1016/j.jhep.2018.05.024. Epub 2018 Jul 1. PMID 30104154
- [Background] Lemoine M, Shimakawa Y, Nayagam S, Khalil M, Suso P, Lloyd J, Goldin R, Njai HF, Ndow G, Taal M, Cooke G, D'Alessandro U, Vray M, Mbaye PS, Njie R, Mallet V, Thursz M. The gamma-glutamyl transpeptidase to platelet ratio (GPR) predicts significant liver fibrosis and cirrhosis in patients with chronic HBV infection in West Africa. Gut. 2016 Aug;65(8):1369-76. doi: 10.1136/gutjnl-2015-309260. Epub 2015 Jun 24. PMID 26109530
- [Background] Shimakawa Y, Lemoine M, Bottomley C, Njai HF, Ndow G, Jatta A, Tamba S, Bojang L, Taal M, Nyan O, D'Alessandro U, Njie R, Thursz M, Hall AJ. Birth order and risk of hepatocellular carcinoma in chronic carriers of hepatitis B virus: a case-control study in The Gambia. Liver Int. 2015 Oct;35(10):2318-26. doi: 10.1111/liv.12814. Epub 2015 Mar 11. PMID 25728498
- [Background] Njai HF, Shimakawa Y, Sanneh B, Ferguson L, Ndow G, Mendy M, Sow A, Lo G, Toure-Kane C, Tanaka J, Taal M, D'alessandro U, Njie R, Thursz M, Lemoine M. Validation of rapid point-of-care (POC) tests for detection of hepatitis B surface antigen in field and laboratory settings in the Gambia, Western Africa. J Clin Microbiol. 2015 Apr;53(4):1156-63. doi: 10.1128/JCM.02980-14. Epub 2015 Jan 28. PMID 25631805
- [Background] Shimakawa Y, Lemoine M, Njai HF, Bottomley C, Ndow G, Goldin RD, Jatta A, Jeng-Barry A, Wegmuller R, Moore SE, Baldeh I, Taal M, D'Alessandro U, Whittle H, Njie R, Thursz M, Mendy M. Natural history of chronic HBV infection in West Africa: a longitudinal population-based study from The Gambia. Gut. 2016 Dec;65(12):2007-2016. doi: 10.1136/gutjnl-2015-309892. Epub 2015 Jul 16. PMID 26185161
- [Background] Shimakawa Y, Lemoine M, Mendy M, Njai HF, D'Alessandro U, Hall A, Thursz M, Njie R. Population-based interventions to reduce the public health burden related with hepatitis B virus infection in the gambia, west Africa. Trop Med Health. 2014 Jun;42(2 Suppl):59-64. doi: 10.2149/tmh.2014-S08. PMID 25425952
- [Derived] Shimakawa Y, Takao Y, Anderson ST, Taal M, Yamaguchi T, Giana L, Ndow G, Sarr L, Kambi A, Njai HF, Bottomley C, Nyan O, Sabally S, D'Alessandro U, Taylor-Robinson SD, Thursz M, Lemoine M, Njie R. The prevalence and burden of symptoms in patients with chronic liver diseases in The Gambia, West Africa. Palliat Med. 2015 Feb;29(2):184-5. doi: 10.1177/0269216314547103. Epub 2014 Sep 5. No abstract available. PMID 25193933